CLINICAL TRIAL: NCT01454661
Title: Probiotic Modulation of Early Microbial Contact in Premature Infants
Brief Title: Probiotics and Early Microbial Contact in Preterm Neonates
Acronym: ProPre
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Samuli Rautava, Principal Investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ETMK 104/180/2011
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Premature; Infant, Light-for-dates; Breastfeeding
Keywords: Probiotics; Premature infant; Intestinal microbiota; Intestinal immunity; Breastfeeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo mother - LGG infant (Active Comparator): Placebo is administered to the lactating mother whilst the infant receives the probiotic LGG.
  Interventions: Dietary Supplement: LGG
- placebo mother - placebo infant (Placebo Comparator): Placebo is administered to both the lactating mother and her infant.
  Interventions: Dietary Supplement: Placebo
- LGG mother - placebo infant (Active Comparator): The probiotic LGG is administered to the lactating mother whilst the infant receives placebo.
  Interventions: Dietary Supplement: LGG
- LGG+Bb-12 mother - Placebo infant (Active Comparator): A combination of the probiotics LGG and Bb-12 is administered to the lactating mother, the infant receives placebo.
  Interventions: Dietary Supplement: LGG+Bb-12
- Pacebo mother - LGG+Bb-12 infant (Active Comparator): Placebo is administered to the lactating mother, the infant receives a combination of the probiotics LGG and Bb-12
  Interventions: Dietary Supplement: LGG+Bb-12

INTERVENTIONS:
Dietary Supplement: LGG — Lactobacillus rhamnosus GG 10E9 cfu / day
  Arms: LGG mother - placebo infant; placebo mother - LGG infant
Dietary Supplement: LGG+Bb-12 — A combination of the probiotics Lactobacillus rhamnosus GG and Bifidobacterium lactis Bb-12 administered 10E9 cfu / day each.
  Arms: LGG+Bb-12 mother - Placebo infant; Pacebo mother - LGG+Bb-12 infant
Dietary Supplement: Placebo — Microcrystalline cellulose is used as placebo.
  Arms: placebo mother - placebo infant

SUMMARY:
Probiotics are live microbes which, when administered in sufficient amounts, confer a health benefit to the host. According to recent clinical trials, administration of probiotics to very low birth weight infants significantly reduces overall mortality and risk of necrotizing enterocolitis, a devastating inflammatory intestinal disease. The investigators have previously demonstrated that administering probiotics to the lactating mother enhances the immunoprotective properties of breast milk. Despite the promising data, the optimal probiotic intervention is yet to be established. The mechanisms by which probiotics exert their effects remain largely unknown.

This research project is based on the notion that modulation of early microbial contact by probiotics may provide a safe and effective means to improve the health of preterm infants. In particular, the investigators hypothesize that the protective potential of probiotics may be enhanced via breast milk by administering probiotics to the lactating mother. All of the potentially beneficial effects of probiotic bacteria are strain-specific and therefore preliminary laboratory and clinical research with regard to different physiological targets of probiotic intervention should be carried out to guide the design of large-scale clinical trials aiming show clinical efficacy and establish clinical practice. The purpose of this research project is to identify targets for probiotic therapy in premature neonates and to provide insight into the optimal probiotic strains and administration protocol the clinical efficacy of which will subsequently be tested in a randomized controlled trial.

The specific aims of the project are:

1. To determine the effect of maternal consumption of probiotics during lactation on immunomodulatory properties of breast milk in mothers of premature infants. Concentrations of immunomodulatory factors and microbiological properties of breast milk will be measured.
2. To investigate the impact of different probiotic administration protocols on gut microbiota composition in preterm infants. In particular, the issue whether maternal probiotic consumption instead or in addition to probiotics administered to the infant is effective will be elucidated. Different potential probiotic strains will be assessed.
3. To elucidate the impact probiotic bacteria administered to the lactating mother and/or directly to the infant on gut immunophysiology in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* premature infant born at <35 weeks gestational age

Exclusion Criteria:

* severe asphyxia
* significant anomalies

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | 1 month
  Assessment of indigenous intestinal microbiota composition in premature neonates during the first month of life

SECONDARY OUTCOMES:
Intestinal immunity | 1 month
  Intestinal immune gene expression profiles will be assessed from fecal samples.
Breast milk compostion | 1 months
  Immunological and microbiological properties of breast milk will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Samuli Rautava, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland